CLINICAL TRIAL: NCT05802121
Title: The Role of Akkermansia Muciniphilia in Combating the Metabolic Effects of Androgen Deprivation Therapy in Men With Metastatic Prostate Cancer
Brief Title: Akkermansia Muciniphilia and Metabolic Side Effects of ADT
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Western University (Other)
Responsible Party: Principal Investigator, Melissa Huynh, Assistant Professor, Western University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ReDA ID 12558
Record Dates: First submitted 2023-03-12; First posted 2023-04-06 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Metabolic Syndrome; Obesity; Cardiovascular Morbidity; Bone Diseases; Hyperlipidemias; Diabetes
Keywords: prostate cancer; metabolic syndrome; androgen deprivation therapy; microbiome; Akkermansias muciniphilia; cardiovascular disease
MeSH Terms: conditions — Prostatic Neoplasms; Metabolic Syndrome; Obesity; Bone Diseases; Hyperlipidemias; Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: This will be a single-institution, randomized controlled trial involving men ≥18 years of age with metastatic castration-sensitive prostate cancer. This study will require histologic confirmation of prostate adenocarcinoma and radiographic evidence of metastatic disease on either conventional imaging (CT and BS) or PSMA PET scan. Patients will be randomized 1:1 to receive acetate supplementation or observation. Our institution sees approximately 200 new metastatic prostate cancer patients each year, therefore, the investigators do not anticipate encountering difficulties with recruitment into this study over a period of 2 years.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apple Cider Vinegar (Experimental): Jamison apple cider vinegar caplets (NPN: 80078433). Each patient will be instructed to take 1 acetate caplet (equivalent of 143 mg/caplet containing 36% acetic acid) per day for 3 months.
  Interventions: Drug: Apple Cider Vinegar
- Observation (No Intervention): Observation group will follow standard of care treatment.

INTERVENTIONS:
Drug: Apple Cider Vinegar — Each patient will be instructed to take 1 caplet (equivalent of 143 mg/caplet containing 36% acetic acid) per day for 3 months (NPN: 80078433)
  https://www.jamiesonvitamins.com/products/apple-cider-vinegar-chromium?srsltid=AfmBOoqdVBFe83_5JM9BmkomQM1LqsJYSFTiP_78cnmehfzVg-4T4Z6o
  Arms: Apple Cider Vinegar

SUMMARY:
The overriding objectives of this study are:

1. Primary outcomes:

   1. To confirm that administration of oral acetate increases the proportion of A. muciniphilia in the stool samples of patients with metastatic, castration-sensitive prostate cancer compared to a standard of care arm.
   2. To confirm tolerability and assess for side effects of oral acetate supplementation.
2. Secondary outcomes:

   1. To determine if increased counts of A. muciniphilia correlate with improved metabolic parameters and improved bone health.

ELIGIBILITY:
For inclusion in this study, patients must fulfill all of the following criteria:

1. Men ≥18 years of age with histologically-proven metastatic castration-sensitive prostate adenocarcinoma planned to receive ADT (TNM stage Tany, Nany, M1) (see Appendix I).
2. Must have baseline imaging with 1) CT of the abdomen, and pelvis and bone scan or 2) PSMA PET scan

Patients fulfilling any of the following criteria are NOT eligible for participation in this study:

1. Age less than 18
2. Primary neuroendocrine prostate cancer
3. Treatment with ADT within the year leading up to enrolment
4. Planned or concurrent use of chromium supplementation for the study duration
5. Planned or concurrent use of apple cider vinegar supplementation for the study duration
6. Unable to provide informed consent or unable to understand or read the English language (unless accompanied by an interpreter)
7. Inadequate liver function (>2x upper limit of normal)
8. Any other condition, chronic disease, or lifestyle factor, that, in the opinion of the Qualified Investigator, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant
9. Use of antibiotics that cannot be discontinued for a washout period and remain off them for the duration of the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Fecal Akkermansia muciniphilia counts | 1 week
  Counts of Akkermansia muciniphilia in participant stool samples at 1 week following the intervention will be compared to baseline counts.
Fecal Akkermansia muciniphilia counts | 1 month
  Counts of Akkermansia muciniphilia in participant stool samples at 1 month following the intervention will be compared to baseline counts.
Fecal Akkermansia muciniphilia counts | 3 month
  Counts of Akkermansia muciniphilia in participant stool samples at 3 months following the intervention will be compared to baseline counts.
Fecal Akkermansia muciniphilia counts | 4 month
  Counts of Akkermansia muciniphilia in participant stool samples at 4 months following the intervention will be compared to baseline counts.
Fecal Akkermansia muciniphilia counts | 6 month
  Counts of Akkermansia muciniphilia in participant stool samples at 6 months following the intervention will be compared to baseline counts.
Side effects and tolerability | 3 months
  We will record side effects reported by the participants and the rate of Discontinuation of the intervention.

SECONDARY OUTCOMES:
Metabolic parameters: fasting plasma glucose | 3 months
  Fasting plasma glucose (mmol/L)
Metabolic parameters: fasting plasma glucose | 6 months
  Fasting plasma glucose (mmol/L)
Metabolic parameters: HbA1C | 3 months
  HbA1c (%)
Metabolic parameters: HbA1c | 6 months
  HbA1c (%)
Metabolic parameters: triglycerides | 3 months
  Triglycerides (mmol/L)
Metabolic parameters: triglycerides | 6 months
  Triglycerides (mmol/L)
Metabolic parameters: LDL cholesterol | 3 months
  LDL cholesterol (mmol/L)
Metabolic parameters: LDL cholesterol | 6 months
  LDL cholesterol (mmol/L)
Metabolic parameters: HDL cholesterol | 3 months
  HDL cholesterol (mmol/L)
Metabolic parameters: HDL cholesterol | 6 months
  HDL cholesterol (mmol/L)
Metabolic parameters: total cholesterol | 3 months
  Total cholesterol (mmol/L)
Metabolic parameters: total cholesterol | 6 months
  Total cholesterol (mmol/L)
Metabolic parameters: PSA | 6 months
  PSA (ng/mL)
Metabolic parameters: PSA | 3 months
  PSA (ng/mL)
Metabolic parameters: hemoglobin | 3 months
  Hemoglobin (g/L)
Metabolic parameters: hemoglobin | 6 months
  Hemoglobin (g/L)
Metabolic parameters: serum creatinine | 3 months
  Serum creatinine (µmol/L)
Metabolic parameters: serum calcium | 3 months
  Serum calcium (µmol/L)
Metabolic parameters: serum calcium | 6 months
  Serum calcium (µmol/L)
Metabolic parameters: alanine transferase | 3 months
  Alanine transferase (U/L)
Metabolic parameters: alanine transferase | 6 months
  Alanine transferase (U/L)
Metabolic parameters: aspartate aminotransferase | 3 months
  Aspartate aminotransferase (U/L)
Metabolic parameters: aspartate aminotransferase | 6 months
  Aspartate aminotransferase (U/L)
Metabolic parameters: Insulin resistance index (HOMA IR) | 3 months
  Insulin resistance index (HOMA IR)
Metabolic parameters: HOMA IR | 6 months
  Insulin resistance index (HOMA IR)
Bone health: dp-ucMGP levels | 3 months
  Circulating plasma dp-ucMGP levels (surrogate for vitamin K2 levels) from baseline
Bone health: dp-ucMGP levels | 6 months
  Circulating plasma dp-ucMGP levels (surrogate for vitamin K2 levels) from baseline
Bone health: Vitamin K2 | 3 months
  Vitamin K2 levels
Bone health: Vitamin K2 | 6 months
  Vitamin K2 levels

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Huynh, MD, Principal Investigator — Western University
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Our study protocol and analyses can be shared, but individual data will not.

REFERENCES:
- [Background] McKay RR, Feng FY, Wang AY, Wallis CJD, Moses KA. Recent Advances in the Management of High-Risk Localized Prostate Cancer: Local Therapy, Systemic Therapy, and Biomarkers to Guide Treatment Decisions. Am Soc Clin Oncol Educ Book. 2020 May;40:1-12. doi: 10.1200/EDBK_279459. PMID 32412803
- [Background] Smith MR, Finkelstein JS, McGovern FJ, Zietman AL, Fallon MA, Schoenfeld DA, Kantoff PW. Changes in body composition during androgen deprivation therapy for prostate cancer. J Clin Endocrinol Metab. 2002 Feb;87(2):599-603. doi: 10.1210/jcem.87.2.8299. PMID 11836291
- [Background] Timilshina N, Breunis H, Alibhai SM. Impact of androgen deprivation therapy on weight gain differs by age in men with nonmetastatic prostate cancer. J Urol. 2012 Dec;188(6):2183-8. doi: 10.1016/j.juro.2012.08.018. Epub 2012 Oct 18. PMID 23083859
- [Background] Braga-Basaria M, Dobs AS, Muller DC, Carducci MA, John M, Egan J, Basaria S. Metabolic syndrome in men with prostate cancer undergoing long-term androgen-deprivation therapy. J Clin Oncol. 2006 Aug 20;24(24):3979-83. doi: 10.1200/JCO.2006.05.9741. PMID 16921050
- [Background] Seible DM, Gu X, Hyatt AS, Beard CJ, Choueiri TK, Efstathiou JA, Miyamoto DT, Mitin T, Martin NE, Sweeney CJ, Trinh QD, Beckman JA, Basaria S, Nguyen PL. Weight gain on androgen deprivation therapy: which patients are at highest risk? Urology. 2014 Jun;83(6):1316-21. doi: 10.1016/j.urology.2014.02.006. Epub 2014 Apr 13. PMID 24726149
- [Background] Sturgeon KM, Deng L, Bluethmann SM, Zhou S, Trifiletti DM, Jiang C, Kelly SP, Zaorsky NG. A population-based study of cardiovascular disease mortality risk in US cancer patients. Eur Heart J. 2019 Dec 21;40(48):3889-3897. doi: 10.1093/eurheartj/ehz766. PMID 31761945
- [Background] Saigal CS, Gore JL, Krupski TL, Hanley J, Schonlau M, Litwin MS; Urologic Diseases in America Project. Androgen deprivation therapy increases cardiovascular morbidity in men with prostate cancer. Cancer. 2007 Oct 1;110(7):1493-500. doi: 10.1002/cncr.22933. PMID 17657815
- [Background] Keating NL, O'Malley AJ, Smith MR. Diabetes and cardiovascular disease during androgen deprivation therapy for prostate cancer. J Clin Oncol. 2006 Sep 20;24(27):4448-56. doi: 10.1200/JCO.2006.06.2497. PMID 16983113
- [Background] Jespersen CG, Norgaard M, Borre M. Androgen-deprivation therapy in treatment of prostate cancer and risk of myocardial infarction and stroke: a nationwide Danish population-based cohort study. Eur Urol. 2014 Apr;65(4):704-9. doi: 10.1016/j.eururo.2013.02.002. Epub 2013 Feb 12. PMID 23433805
- [Background] D'Amico AV, Denham JW, Crook J, Chen MH, Goldhaber SZ, Lamb DS, Joseph D, Tai KH, Malone S, Ludgate C, Steigler A, Kantoff PW. Influence of androgen suppression therapy for prostate cancer on the frequency and timing of fatal myocardial infarctions. J Clin Oncol. 2007 Jun 10;25(17):2420-5. doi: 10.1200/JCO.2006.09.3369. PMID 17557956
- [Background] Voog JC, Paulus R, Shipley WU, Smith MR, McGowan DG, Jones CU, Bahary JP, Zeitzer KL, Souhami L, Leibenhaut MH, Rotman M, Husain SM, Gore E, Raben A, Chafe S, Sandler HM, Efstathiou JA. Cardiovascular Mortality Following Short-term Androgen Deprivation in Clinically Localized Prostate Cancer: An Analysis of RTOG 94-08. Eur Urol. 2016 Feb;69(2):204-10. doi: 10.1016/j.eururo.2015.08.027. Epub 2015 Sep 9. PMID 26362090
- [Background] Efstathiou JA, Bae K, Shipley WU, Hanks GE, Pilepich MV, Sandler HM, Smith MR. Cardiovascular mortality after androgen deprivation therapy for locally advanced prostate cancer: RTOG 85-31. J Clin Oncol. 2009 Jan 1;27(1):92-9. doi: 10.1200/JCO.2007.12.3752. Epub 2008 Dec 1. PMID 19047297
- [Background] Grossmann M, Hamilton EJ, Gilfillan C, Bolton D, Joon DL, Zajac JD. Bone and metabolic health in patients with non-metastatic prostate cancer who are receiving androgen deprivation therapy. Med J Aust. 2011 Mar 21;194(6):301-6. doi: 10.5694/j.1326-5377.2011.tb02979.x. PMID 21426285
- [Background] Morote J, Orsola A, Abascal JM, Planas J, Trilla E, Raventos CX, Cecchini L, Encabo G, Reventos J. Bone mineral density changes in patients with prostate cancer during the first 2 years of androgen suppression. J Urol. 2006 May;175(5):1679-83; discussion 1683. doi: 10.1016/S0022-5347(05)00999-7. PMID 16600728
- [Background] Smith MR, Lee WC, Brandman J, Wang Q, Botteman M, Pashos CL. Gonadotropin-releasing hormone agonists and fracture risk: a claims-based cohort study of men with nonmetastatic prostate cancer. J Clin Oncol. 2005 Nov 1;23(31):7897-903. doi: 10.1200/JCO.2004.00.6908. PMID 16258089
- [Background] Kokorovic A, So AI, Serag H, French C, Hamilton RJ, Izard JP, Nayak JG, Pouliot F, Saad F, Shayegan B, Aprikian A, Rendon RA. Canadian Urological Association guideline on androgen deprivation therapy: Adverse events and management strategies. Can Urol Assoc J. 2021 Jun;15(6):E307-E322. doi: 10.5489/cuaj.7355. No abstract available. PMID 34127184
- [Background] Daisley BA, Chanyi RM, Abdur-Rashid K, Al KF, Gibbons S, Chmiel JA, Wilcox H, Reid G, Anderson A, Dewar M, Nair SM, Chin J, Burton JP. Abiraterone acetate preferentially enriches for the gut commensal Akkermansia muciniphila in castrate-resistant prostate cancer patients. Nat Commun. 2020 Sep 24;11(1):4822. doi: 10.1038/s41467-020-18649-5. PMID 32973149
- [Background] van der Beek CM, Canfora EE, Lenaerts K, Troost FJ, Damink SWMO, Holst JJ, Masclee AAM, Dejong CHC, Blaak EE. Distal, not proximal, colonic acetate infusions promote fat oxidation and improve metabolic markers in overweight/obese men. Clin Sci (Lond). 2016 Nov 1;130(22):2073-2082. doi: 10.1042/CS20160263. Epub 2016 Jul 20. PMID 27439969
- [Background] Everard A, Belzer C, Geurts L, Ouwerkerk JP, Druart C, Bindels LB, Guiot Y, Derrien M, Muccioli GG, Delzenne NM, de Vos WM, Cani PD. Cross-talk between Akkermansia muciniphila and intestinal epithelium controls diet-induced obesity. Proc Natl Acad Sci U S A. 2013 May 28;110(22):9066-71. doi: 10.1073/pnas.1219451110. Epub 2013 May 13. PMID 23671105
- [Background] Perraudeau F, McMurdie P, Bullard J, Cheng A, Cutcliffe C, Deo A, Eid J, Gines J, Iyer M, Justice N, Loo WT, Nemchek M, Schicklberger M, Souza M, Stoneburner B, Tyagi S, Kolterman O. Improvements to postprandial glucose control in subjects with type 2 diabetes: a multicenter, double blind, randomized placebo-controlled trial of a novel probiotic formulation. BMJ Open Diabetes Res Care. 2020 Jul;8(1):e001319. doi: 10.1136/bmjdrc-2020-001319. PMID 32675291
- [Background] Zhou Q, Zhang Y, Wang X, Yang R, Zhu X, Zhang Y, Chen C, Yuan H, Yang Z, Sun L. Gut bacteria Akkermansia is associated with reduced risk of obesity: evidence from the American Gut Project. Nutr Metab (Lond). 2020 Oct 22;17:90. doi: 10.1186/s12986-020-00516-1. eCollection 2020. PMID 33110437
- [Background] Luna M, Guss JD, Vasquez-Bolanos LS, Castaneda M, Rojas MV, Strong JM, Alabi DA, Dornevil SD, Nixon JC, Taylor EA, Donnelly E, Fu X, Shea MK, Booth SL, Bicalho R, Hernandez CJ. Components of the Gut Microbiome That Influence Bone Tissue-Level Strength. J Bone Miner Res. 2021 Sep;36(9):1823-1834. doi: 10.1002/jbmr.4341. Epub 2021 Jun 4. PMID 33999456
- [Background] Booth SL, Tucker KL, Chen H, Hannan MT, Gagnon DR, Cupples LA, Wilson PW, Ordovas J, Schaefer EJ, Dawson-Hughes B, Kiel DP. Dietary vitamin K intakes are associated with hip fracture but not with bone mineral density in elderly men and women. Am J Clin Nutr. 2000 May;71(5):1201-8. doi: 10.1093/ajcn/71.5.1201. PMID 10799384
- [Background] Evenepoel P, Dejongh S, Verbeke K, Meijers B. The Role of Gut Dysbiosis in the Bone-Vascular Axis in Chronic Kidney Disease. Toxins (Basel). 2020 Apr 29;12(5):285. doi: 10.3390/toxins12050285. PMID 32365480
- [Background] Mandatori D, Pelusi L, Schiavone V, Pipino C, Di Pietro N, Pandolfi A. The Dual Role of Vitamin K2 in "Bone-Vascular Crosstalk": Opposite Effects on Bone Loss and Vascular Calcification. Nutrients. 2021 Apr 7;13(4):1222. doi: 10.3390/nu13041222. PMID 33917175
- [Background] Arrieta MC, Bistritz L, Meddings JB. Alterations in intestinal permeability. Gut. 2006 Oct;55(10):1512-20. doi: 10.1136/gut.2005.085373. No abstract available. PMID 16966705